CLINICAL TRIAL: NCT06755450
Title: A Phase 1, Open Label, Dose Escalation, Multicenter, First-in-Human (FIH) Study Evaluating the Safety, Pharmacokinetics and Pharmacodynamics of Oral AUR112 In Patients With Relapsed Advanced Lymphoma (ADITI-1)
Brief Title: Study Evaluating Safety Pharmacokinetics and Pharmacodynamics of AUR112 in Patients With Relapsed Advanced Lymphoma
Acronym: ADITI-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aurigene Discovery Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AUR112-101
Record Dates: First submitted 2024-12-31; First posted 2025-01-01 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Advanced Lymphomas
Keywords: Non-Hodgkin Lymphoma (NHL); Hodgkin Lymphoma; Relapse Advanced Lymphomas
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Intervention Model Description: Sequential Assignment Dose Escalation Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUR112 (Experimental): Experimental: AUR112, 100mg to 1200mg Currently, six (6) planned dose levels are 100 mg, 200 mg, 400 mg, 600 mg, 900 mg, and 1200 mg once daily (QD).
  AUR112: Once daily
  Interventions: Drug: AUR112

INTERVENTIONS:
Drug: AUR112 — Once daily

SUMMARY:
A Phase 1, Open Label, Dose Escalation, Multicenter, First-in-Human (FIH) Study Evaluating the Safety, Pharmacokinetics and Pharmacodynamics of Oral AUR112 in Patients with Relapsed Advanced Lymphoma (ADITI-1)

DETAILED DESCRIPTION:
The main objective of Part 1 will be to evaluate the safety and tolerability of the study drug AUR112.

Dose escalation of single agent AUR112 will be conducted in the classic 3+3 design. Safety including Dose Limiting Toxicities (DLTs), PK, and PD will be assessed at each dose. Dose escalation will continue until safety limits are reached or the escalation will stop earlier if PK/PD data suggest that a biologically active dose has reached.

The objective is to determine dose(s) which will be investigated in future trials.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age
2. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
3. Acceptable bone marrow and organ function at screening as described below:

   1. ANC ≥ 1000/μL (without WBC growth factor support)
   2. Platelet count: For patients with CLL ≥ 50,000/μL; For patients with lymphomas ≥ 75,000/μL without bone marrow involvement and ≥ 50,000/μL with bone marrow involvement. These thresholds should be qualified without platelet transfusion support.
   3. Hemoglobin ≥ 9 g/dL (RBC Transfusion is allowed to achieve this Hb)
   4. Total Bilirubin ≤ 1.5 x ULN; (Patients with known Gilbert's syndrome are allowed with a Total Bilirubin ≤ 2.5 x ULN)
   5. AST (SGOT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases)
   6. ALT (SGPT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases)
   7. Creatinine clearance (CrCl) ≥ 60 mL/min (either measured or estimated by the Cockcroft-Gault formula). (Cockcroft-Gault formula for estimated creatinine clearance [eCrCl]: eCrCl = [140- Age] × Weight [kg] × [0.85 if Female] / [72 × serum creatinine (mg/dL)]).
4. Ability to swallow and retain oral medications
5. Histopathological diagnosis of Non-Hodgkin Lymphoma (NHL) or Chronic Lymphocytic Leukemia (CLL) or Hodgkin disease. Note:

5a. The lymphoma should be either in Stage III or IV according to Lugano classification (Cheson et al. 2014) at screening. 5b. The lymphomas included in this study must fall within one of the following 2017 World Health Organization categories except lymphoma mentioned in Exclusion criterion #5:

* Mature B-cell neoplasms (excluding plasma cell neoplasms, heavy chain disease, and primary central nervous system [CNS] lymphoma).
* Mature T- and NK-cell neoplasms.
* Hodgkin lymphomas 5c. The CLL should be Binet Stage C/Rai stage III or IV, as per the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines (Hallek et al. 2018).

  6. In the case of subjects who have lymphoma for which high-dose chemotherapy and autologous stem cell transplantation (HDASCT) is considered a standard curative therapy, eligibility for this study requires that the subject's disease has relapsed after HDASCT, or the subject is not eligible for HD-ASCT, or that the subject has refused HD-ASCT.

  7. In the case of patients who have lymphoid malignancies for which CAR-T therapy is indicated, eligibility for this study requires that the disease has relapsed after CAR-T, or the patient is not eligible for CAR-T, or the patient has refused CAR-T, or the CAR-T is not available locally.

  8. Evidence of measurable disease as per Lugano Criteria for Lymphoma (Cheson et al. 2014) or evidence of measurable disease as per iwCLL Criteria for CLL (Hallek et al. 2018). Note: Patients with Small Lymphocytic Lymphoma (SLL) alone or in combination with CLL are allowed.

  9. Standard curative measures do not exist, and the patient must have exhausted all effective therapies available locally. The patients must have relapsed or refractory to at least 2 prior lines of systemic therapies for NHL or CLL, or Hodgkin disease.

Note:

* Any cancer patient with access to any effective therapy locally must not be enrolled.
* Patients with CLL should have documented evidence for progressive or symptomatic disease (active disease) and must have indications for treatment (Hallek et al 2018).
* Patients with indolent lymphomas also must have indications for treatment, such as the GELF (Brice et al 1997) or BNLI criterion (Ardeshna et al 2003)

Exclusion Criteria:

1. Systemic anti-cancer therapy, such as chemotherapy, biological therapy, or immunomodulatory drug therapy received within the past 28 days or 5 half-lives, whichever is longer, from the Cycle 1 Day 1 of the study. Note: Concomitant use of low dose prednisone (up to 10 mg/day) is allowed
2. Presence of an acute or chronic toxicity resulting from prior anticancer treatment, with the exception of alopecia or nail changes, that has not resolved to Grade ≤ 1, as determined by NCI CTCAE v 5.0. 1
3. Definitive Radiotherapy within the last 21 days of Cycle 1 Day 1 (limited field palliative radiation is allowed and no restrictions during the screening period or during the trial).
4. Use of any investigational agent within 28 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1
5. Patients with Burkitt's lymphoma, Burkitt-like lymphoma, posttransplant lymphoproliferative disease, primary mediastinal large-B cell lymphoma, cutaneous lymphomas, mycosis fungoides (MF), or Sezary syndrome (SS).
6. Known symptomatic or untreated or recently treated (≤ 6 months of screening) central nervous system (CNS) lymphoma. Patients with previously treated (> 6 months of screening) CNS lymphoma and are now stable and asymptomatic, from CNS perspective, are allowed.
7. Patients with lymphoma that requires immediate cytoreductive therapy.
8. Patients with low-grade lymphoma or indolent lymphoma that does not meet conventional criteria (Jeong SH, 2022) for requiring treatment.
9. Patients on drugs which are inhibitors of P-gp or BCRP or UGT1A1 and when these drugs cannot be discontinued from at least one week prior to Cycle 1 Day 1. Note: These drugs will be prohibited during Cycle 1 of therapy.
10. Major surgery ≤ 28 days from Cycle 1 Day 1 (major surgery is defined as a procedure requiring general anesthesia)
11. Active infection requiring systemic therapy. Note: Prophylactic use of antibiotics is allowed. Any infection detected during screening period which is resolved adequately according to investigator before the Cycle 1 Day 1, is allowed.
12. Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome-related illness.
13. Known active or chronic hepatitis B (HBsAg +ve) or hepatitis C infection (HCV antibody +ve).
14. The patient who is expected to require any other form of antineoplastic therapy or targeted therapy while on study
15. . Uncontrolled congestive heart failure (New York Heart Association [NYHA] Class 2-4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, or transient ischemic attack, or pulmonary embolism within 3 months prior to Cycle 1 Day 1.
16. Ongoing cardiac dysrhythmias requiring treatment of any grade or treatment of cardiac dysrhythmias in past 3 months, before Cycle 1 Day 1.
17. QTcF (Fridericia) interval >470 ms on ECG at screening and/or at Cycle 1 Day 1 pre-dose.
18. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or significant gastritis, active bleeding diatheses, presence of any major medical illness (e.g. renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, or psychiatric illness/social situations or clinically significant laboratory / ECG abnormalities at screening, any or a combination of illnesses, which, in the opinion of the PI, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
19. Current swab-positive or suspected (under investigation) Covid19 infection or fever and other signs or symptoms suggestive of Covid-19 infection with recent contact of person(s) with confirmed Covid-19 infection, at screening or Cycle 1 Day 1.
20. History of another primary malignancy within 5 years prior to starting study drug, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study.
21. Positive pregnancy test for women of child-bearing potential (WOCBP) at the screening or enrolment visit.
22. Lactating women or WOCBP or a man with a partner who has childbearing potential, who are neither surgically sterilized nor willing to use reliable contraceptive methods(hormonal contraceptive, IUD, or any double combination of male or female condom, spermicidal gel, diaphragm, sponge, cervical cap) during the screening period, while on AUR112 and at least 28 days after last dose

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
First cycle Dose Limiting Toxicities (DLT). | 28 days (Cycle 1)
  Number of participants with dose limiting toxicities (DLT) taking AUR112
Safety of AUR112 as measured by the number of participants with treatment related adverse events (AE) graded according to NCI CTCAE version 5.0 | 28 days
  The assessment of safety was based on the frequency of deaths, adverse event (AE), serious adverse event (SAE)s leading to discontinuation of study drug, and abnormalities in specific laboratory assessments. AEs and laboratory values will be graded for severity according to NCI CTCAE version 5.0
To determine the doses to be recommended for evaluation in future studies. | 28 days
  Determine selected dose(s) to be studied in future clinical trials
Pharmacokinetics: Maximum concentration (Cmax) | [Time Frame: Day 1 and Day 15]
  Maximum concentration of AUR112
Pharmacokinetics: Time to Maximum concentration (Tmax) | [Time Frame: Day 1 and Day 15]
  Tmax in hours
Pharmacokinetics: Area under the curve (AUC) | [Time Frame: Day 1 and Day 15]
  Area under the curve (AUC) of AUR 112 in h* mcg/mL
Pharmacokinetics: Mean Residence Time (MRT) | [Time Frame: Day 1 and Day 15]
  Average time the drugs stays in the body
Pharmacokinetics: Terminal elimination half-life | [Time Frame: Day 1 and Day 15]
  Terminal elimination half-life of AUR 112 in hours
Maximum concentration (Cmax) administered under fasting/fed condition | [Time Frame: Day 8 and Day 9]
  Compare in fast and fed conditions
Time to Maximum concentration (Tmax) administered under fasting/fed condition | [Time Frame: Day 8 and Day 9]
  Compare Tmax in fast and fed conditions
Area under curve (AUC) administered under fasting/fed condition | [Time Frame: Day 8 and Day 9]
  Compare AUC in fast and fed conditions

OTHER OUTCOMES:
Exploratory endpoint: Expression of cytokines | [Time Frame: Day 1, Day 2, and Day 15]
  Pharmacodynamic marker: CYTOKINE MARKERS analysis
Exploratory endpoint: Gene expression profile | [Time Frame: Day 1, Day 2, and Day 15]
  Pharmacodynamic marker: Gene expression analysed from whole blood
Exploratory endpoint- Efficacy assessments, Overall Response Rate | [Time Frame: Through study completion, an average of 1 year]
  Efficacy assessments-Overall Response Rate
Exploratory endpoint- Efficacy assessments, Duration of Response | [Time Frame: Through study completion, an average of 1 year]
  Efficacy assessments- Duration of Response
Exploratory endpoint- Efficacy assessments, Progression Free Survival (PFS) | [Time Frame: Through study completion, an average of 1 year]
  Efficacy assessments- Progression Free Survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Kumar, Principal Investigator — Aurigene Oncology Limited
Locations (19):
- India (19):
  - Sir Sayajirao General Hospital (SSG), Vadodara, Gujarat
  - National Cancer Institute , All India Institute of Medical Sciences, Jhajjar, Haryana
  - Health Care Global Enterprises, Bangalore, Karnataka
  - Srinivasam Cancer Care Multi Speciality Hospitals India Pvt Ltd. , Bangalore 560072., Bangalore, Karnataka
  - Jeevan Amrut Hematology Center, Aurangabad, Aurangabad, Maharashtra
  - HCG Cancer Centre, Nagpur, Maharashtra
  - Sahyadri Hospital Private Limited, Pune, Maharashtra
  - Novo Solitaire Care, Pune, Maharashtra
  - Armed Forces Medical College, Pune, Maharashtra
  - Onco Life Cancer, Centre, Satara, Satara, Maharashtra
  - Sunact Cancer Institute Pvt. Ltd, Thane, Maharashtra
  - Siddharth Gupta Memorial Hospital,, Wardha, Maharashtra
  - Tata Memorial Hospital, Pārel, Mumbai
  - AIIMS, New Delhi, New Delhi, New Delhi
  - Max Super Specialty Hospital, Saket, New Delhi
  - AIIMS, Bhubaneswar, Bhubaneswar, Odisha
  - Somani Hospital, Jaipur, Rajasthan
  - AIIMS, Rishikesh, Rishikesh, Uttarakhand
  - Tata Medical Centre, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No